CLINICAL TRIAL: NCT04668417
Title: Patient Portal Reminder/Recall for Influenza Vaccination in the UCLA Health System- Pediatric Second Dose
Brief Title: Pediatric Second Influenza Dose Portal Reminder Recall
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Professor of Pediatrics, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 17-001889-AM-00013; 5R01AI135029 (NIH)
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Influenza; Respiratory Tract Infections
Keywords: Vaccination; Reminder Recall; Patient Portal
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reminders with direct scheduling link (Active Comparator): Patient proxy receives a reminder/recall messages regarding second dose influenza vaccination via the patient portal with a link enabling direct scheduling
  Interventions: Behavioral: Portal Reminders for Second Dose of Influenza Vaccine with Direct Scheduling Link
- Reminders with no direct scheduling link (Active Comparator): Patient proxy receives a reminder/recall messages regarding second dose influenza vaccination via the patient portal with no direct scheduling link
  Interventions: Behavioral: Portal Reminders for Second Dose of Influenza Vaccine without Direct Scheduling Link

INTERVENTIONS:
Behavioral: Portal Reminders for Second Dose of Influenza Vaccine with Direct Scheduling Link — Patient proxy receives reminder/recall messages via the patient portal to get a second dose of influenza vaccine with a direct scheduling link included, enabling the patient to directly schedule a flu vaccination only visit
  Arms: Reminders with direct scheduling link
Behavioral: Portal Reminders for Second Dose of Influenza Vaccine without Direct Scheduling Link — Patient proxy receives reminder/recall messages via the patient portal to get a second dose of influenza vaccine with no direct scheduling link included
  Arms: Reminders with no direct scheduling link

SUMMARY:
This trial is taking place in Los Angeles, CA among patients from primary care practices within the UCLA Health System.

The study design is a parallel 2-arm trial. The parallel arms are 1) a reminder letter for the second dose of influenza vaccine (reminder messages sent via the patient portal) with a direct appointment scheduling link included in the reminder and 2) a reminder letter for the second dose of influenza vaccine, but no direct appointment scheduling link included.

DETAILED DESCRIPTION:
This trial is taking place in Los Angeles, CA among patients from primary care practices within the UCLA Health System, using a parallel 2-arm trial.

Sub-optimal vaccination rates are a significant problem in the U.S., despite their effectiveness in preventing morbidity and mortality from vaccine-preventable illness. In the U.S., annual epidemics of influenza cause substantial morbidity in the U.S. with up to 40,00-80,000 deaths/year and many hospitalizations, emergency and outpatient visits, and significant costs.

Young children-especially those younger than 2- are at high risk of developing serious flu-related complications. Children ages of 6 months to 8 years getting vaccinated for the first time with influenza vaccine should get two doses, and those who have only previously gotten one dose of influenza vaccine, should get a second dose (spaced at least 4 weeks apart).

Reminder/recall (R/R) messages, sent by phone, mail or other modality, can improve child vaccination rates. However, the majority of pediatric or adult primary care practices to not conduct R/R. Barriers are lack of finances, personnel, and algorithms to identify eligible patients. A technological breakthrough that might overcome these barriers involves patient portals-- secure, web-based communication systems, embedded within electronic health records (EHRs), for patients and providers to communicate with each other via email and the internet. Portals are increasingly used by healthcare systems.

This randomized controlled trial will assess the effectiveness of reminders messages, sent to the proxy of pediatric patients ages 6 months to <36 months of age eligible for a second dose of the influenza vaccine based on data in the EHR. Patients will be randomized into one of two arms to receive 1) a reminder letter for a second dose of influenza vaccine, with a direct appointment scheduling link included in the letter or 2) a reminder letter for a second dose of influenza vaccine, without a direct appointment scheduling link included in the letter.

ELIGIBILITY:
Inclusion Criteria:

* Patient within the UCLA Health System identified as a primary care patient per an internal algorithm
* Identified as being overdue for a second dose of influenza vaccine.

Exclusion Criteria:

* Patient within the UCLA Health System not identified as a primary care patient per an internal algorithm
* Not due for a second dose of influenza vaccine.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 698 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Number of patients who received a second dose of influenza vaccine | 3.5 months
  Receipt of a second dose of influenza vaccine (between 12/15/2020 and 4/1/21) among patients. Outcomes will be assessed via vaccine data extraction from the electronic health record and external claims and pharmacy data. The patient must also be an active UCLA Health MyChart user (>= 1 login over the last 12 months from 12/15/2020), excluding activity on the user's initial profile activation date. Individuals not affiliated with any primary care practice will be excluded from the analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Peter G Szilagyi, MD, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California LA, Los Angeles, California, United States